CLINICAL TRIAL: NCT02461706
Title: Physician Expanded Access to Investigational New Drug Cannabidiol for the Treatment of Drug Resistant Epilepsy
Brief Title: Treatment of Drug Resistant Epilepsy
Acronym: Cannabidiol
Status: No longer available | Type: Expanded Access
Sponsor: University of Florida (Other)
Collaborators: James and Esther King Biomedical Research Program (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201401013; FLGV (Other Grant/Funding Number: Florida Department of Health)
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Epilepsy
Keywords: Drug resistant epilepsy
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy | interventions — Cannabidiol; Hematologic Tests

INTERVENTIONS:
Drug: cannabidiol — All subjects will have a dosing titration starting with 25 mg/kg/day and will be titrated weekly as tolerated based on clinical response. All subjects will be clinically evaluated at baseline, once a month for three months and every three months thereafter. In order to ensure safe use at higher doses, patients receiving more than 600 mg of daily CBD will be evaluated at least monthly until they achieve steady state at the final fixed maintenance dose.
  Other Names: CBD
Other: Blood Test — All subjects will have the following clinical laboratory tests including changes in bone marrow (CBC), liver (AST, ALT), and kidney function (creatinine, electrolytes, BUN) will be assessed at baseline, each month during months 1 to 3, and every 3 months thereafter.

SUMMARY:
The main goal of this study is to provide treatment with cannabidiol (CBD) to children with drug resistant epilepsy through a Physician Expanded Access Investigation New Drug protocol. As the controlled therapeutic use of CBD in children is novel, the primary objective of this study is to evaluate the safety and efficacy of CBD when administered as adjunctive therapy in children that have exhausted the majority of FDA approved antiepileptic drug treatment options.

DETAILED DESCRIPTION:
Fifty, (50) children will be provided CBD as part of the Principal Investigator's Physician Expanded Access IND. CBD will be administered as an adjunct to all current antiepileptic drugs. After the screening visit, a 4 week baseline period will be followed and seizures will be recorded in the seizure diary given to the patient at this time. The patients will be clinically evaluated at baseline, once a month for three months and once every three months thereafter. For the first week after study initiation, patients will be called at day 3 to review any changes in condition and again at day 7 to review any changes in condition and to determine whether an increase in dosing is required. Subsequently, patients will be called each week during the titration period to review any changes in condition and determine whether an increase in dosing is required. Maximal dose titration should be achieved in most patients within 5 weeks. In order to ensure safe use at higher doses, patients who receive more than 600 mg of daily CBD will be evaluated at least monthly until they achieve steady state at their final fixed maintenance dose. The investigator will be available by telephone or email throughout the initial four months of the study in between the visits.

ELIGIBILITY:
Inclusion Criteria:

* history of a trial of at least four drugs, including one trial of a combination of two concomitant drugs, without successful seizure control.
* Vagal nerve stimulation: VNS must be on stable settings for a minimum of 1 month,
* RNS deep brain stimulation, or
* the ketogenic diet can be considered equivalent to a drug trial and must be on a stable ratio for a minimum of 3 months.
* anti-epileptic drugs at stable doses for a minimum of 4 weeks prior to enrollment.
* 4 clinically countable seizures per month: Seizure history to include a documented history of generalized seizures (drop attacks, atonic, tonic-clonic and/or myoclonic), focal seizures without loss of consciousness with a motor component, focal seizures with loss of consciousness, or focal seizures with secondary generalization,

Exclusion Criteria:

* Use of CBD based product within the previous 30 days.
* Initiation of felbamate within 6 months.
* Allergy to CBD or any cannabinoid.
* Unable to comply with study visits/requirements.
* Diagnosis of Dravet Syndrome or Lennox-Gastaut syndrome will be excluded completely from this trial.
* Cannabidiol is contraindicated in pregnancy. Female subjects who are pregnant will be excluded from the study. If a female subject is able to become pregnant, she will be given a serum pregnancy test before entry into the study. Female subjects will be informed not become pregnant while taking cannabidiol. Female subjects must tell the investigator and consult an obstetrician or maternal-fetal specialist if they become pregnant during the study.

Ages: 2 Years to 16 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Steven Winesett, MD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Flordia CRC, Gainesville, Florida
  - Nicklaus Children's Hospital, Miami Children's Health System, Miami, Florida